CLINICAL TRIAL: NCT02177747
Title: Comparison of Smartphone-based Ophthalmoscopy Versus Dilated Ophthalmic Examination for Diabetic and Nondiabetic Eye Disease
Brief Title: Smartphone-based Ophthalmoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: Luisa Delcassi (Unknown); Nausica Ghilardi (Unknown)
Responsible Party: Principal Investigator, Andrea Russo, MD, PhD Researcher, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group
Other Study IDs: SMART001
Record Dates: First submitted 2014-06-24; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Diabetic Retinopathy Grading

ARMS (1):
- Diabet patients (Experimental): Smartphone ophthalmoscopy followed by traditional slit-lamp dilated ophthalmoscopy
  Interventions: Other: Ophthalmoscopy conducted using a smartphone equipped with a compact addon; Device: Smartphone

INTERVENTIONS:
Other: Ophthalmoscopy conducted using a smartphone equipped with a compact addon
Device: Smartphone

SUMMARY:
A subset of 120 diabetic patients underwent dilated examination and smartphone ophthalmoscopy. The smartphone was equipped with a compact add-on that filtered and delivered the smartphone's LED light coaxially to the camera, allowing a clear and convenient view of the retina.

ELIGIBILITY:
Inclusion Criteria:

* type 1 or 2 diabetes
* ability to provide written informed consent

Exclusion Criteria:

* significant optic media opacities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Diabetic retinopathy grading | The same day as dilated ophthalmic examination
  The grading was performed according to the Early Treatment Diabetic Retinopathy Study (ETDRS) diabetic retinopathy classification.
  Grade 0: no diabetic retinopathy Grade 1: mild non-proliferative diabetic retinopathy Grade 2: average non-proliferative diabetic retinopathy Grade 3: severe non-proliferative diabetic retinopathy Grade 4: proliferative diabetic retinopathy

CONTACTS AND LOCATIONS:
Locations (1):
- Spedali Civili di Brescia, Brescia, BS, Italy